CLINICAL TRIAL: NCT07043504
Title: Study on the Dynamic Changes of Serum IGF-1 After Cerebral Hemorrhage and Its Correlation With Prognosis of Patients
Brief Title: Study on Dynamic Changes of Serum IGF-1 Post-Cerebral Hemorrhage and Its Prognostic Correlation
Status: Not yet recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yin Yanmei, Yin Yanmei, Shengjing Hospital
Other Study IDs: 2025PS1176K(X1)
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Insulin-Like Growth Factor I
Keywords: Intracerebral Hemorrhage; Prognosis; IGF-1
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to dynamically observe the dynamic changes of serum IGF-1 after intracerebral hemorrhage, explore the impact and correlation of serum IGF-1 with the severity of the patient's condition and prognosis, and provide a reference for clinical treatment timing.

DETAILED DESCRIPTION:
Research Objectives

1. Monitor the dynamic changes in serum IGF-1 concentration in patients with intracerebral hemorrhage at different time points (within 3 days, 14 days, 1 month, 2 months, and 4 months after onset).
2. Analyze the correlation between serum IGF-1 levels and the severity of intracerebral hemorrhage, imaging findings, and prognosis.
3. Explore the clinical value of serum IGF-1 as a biomarker for intracerebral hemorrhage repair.
4. Provide a reference for the clinical treatment timing of IGF-1-related drugs and therapies (such as rh growth hormone, rhIGF-1, etc.).

   Experimental Methods

   Screening Period:

   Within 3 days after onset, record the demographic data, etiology, medical history, complications, disease course, and main clinical manifestations of the subjects during the screening period. Blood sampling for laboratory tests (between 06:00-08:00 in the morning within 3 days after onset) includes: complete blood count, IGF-1, GH, IGFBP-3, LDL-C, thyroid function T4, serum cortisol, ACTH, testosterone or progesterone, serum CRP, fasting blood glucose, glycated hemoglobin. Perform head CT and NIHSS scoring.

   Follow-up Period:

   At the 15th day, 1st month, and 2nd month of the subject's disease course:

   Conduct laboratory tests for IGF-1, GH, and IGFBP-3. Evaluate using the Modified Barthel Index (MBI), Modified Rankin Scale (MRS), Glasgow Coma Scale (GCS), Mini-Mental State Examination (MMSE), PHQ-9 Depression Screening Scale (PHQ-9), and World Health Organization Quality of Life-BREF (WHOQOL-BREF).

   At the 4th month of the subject's disease course:

   Perform laboratory tests for complete blood count, IGF-1, GH, IGFBP-3, LDL-C, thyroid function T4, serum cortisol, ACTH, testosterone or progesterone, CRP, fasting blood glucose, and glycated hemoglobin.

   Evaluate using the same scales as above (MBI, MRS, GCS, MMSE, PHQ-9, WHOQOL-BREF).

   Grouping Based on Dynamic Changes in Serum IGF-1:

   Convert IGF-1 values to IGF-1 SD (standard deviation) by referencing the age-specific reference values for IGF-1 in healthy Chinese populations (Peking Union Medical College).

   IGF-1 Decreased Group: IGF-1 < 0SD IGF-1 Normal Group: 0SD ≤ IGF-1 ≤ 2SD

   Dynamic change-based grouping:

   ① Persistent IGF-1 Decrease Group: IGF-1 remains < 0SD throughout dynamic observation.

   ② IGF-1 Decrease to Normal Group: IGF-1 first < 0SD, then recovers to > 0SD.

   ③ Persistent IGF-1 Normal Group: IGF-1 remains > 0SD throughout dynamic observation.

   Statistical Analysis Based on Experimental Data

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years old;
2. Patients with intracerebral hemorrhage (NIHSS ≥5 points);
3. No history of cerebrovascular diseases with residual functional impairment before brain injury;
4. Hospitalized within 72 hours after injury;
5. BMI ≤28.

Exclusion Criteria:

1. Patients with severe cardiac, hepatic, renal, or pulmonary dysfunction;
2. Glycated hemoglobin >9.0% at screening;
3. History of hypothalamic-pituitary related diseases or severe endocrine diseases;
4. Use of drugs affecting endocrine function (such as glucocorticoids, growth hormones) within the past six months;
5. Pregnant patients. -

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with intracerebral hemorrhage from Shengjing Hospital Affiliated to China Medical University and those from Northern Theater General Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The relationship between serum IGF-1 levels within 3 days after intracerebral hemorrhage and the severity of the condition (referring to NIHSS score) | 3 days after intracerebral
  Serum IGF-1 levels decrease in the acute phase after intracerebral hemorrhage, and the decrease is correlated with the severity of the condition. (The more severe the condition, the larger the number of patients with reduced IGF-1 levels, and the more significant the decrease in IGF-1 values.)，The higher the IGF-1 level, the lower the NIHSS score.

SECONDARY OUTCOMES:
The correlation between the dynamic change trend of IGF-1 after intracerebral hemorrhage and the prognosis of patients | The 5th month
  Patients with persistently decreasing IGF-1 levels have worse functional prognosis than those with persistently normal IGF-1 levels.

IPD SHARING:
Plan to Share IPD: No